CLINICAL TRIAL: NCT01337414
Title: Tools to Optimize Patient Presentation After Onset of Exudative AMD (Using the VMS Interactive Education and Early Detection Multi-Test)
Brief Title: Tools to Optimize Patient Presentation After Onset of Exudative Age-Related Macular Degeneration (AMD)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of financial support
Sponsor: Johns Hopkins University (Other)
Collaborators: Results Group LLC (Industry); National Eye Institute (NEI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: NA_00016895; 2R44EY018990-02 (NIH)
Record Dates: First submitted 2011-04-15; First posted 2011-04-18 (Estimated); Last update posted 2019-08-14 (Actual); Status verified 2019-08

CONDITIONS: Age-related Macular Degeneration
Keywords: age-related macular degeneration; screening; monitoring; diagnosis; dry or non-neovascular age-related macular degeneration (high risk, intermediate, geographic atrophy or AREDS grade 3/4 AMD)
MeSH Terms: conditions — Macular Degeneration; Disease; Geographic Atrophy | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Patient education and self-monitoring vs. customary care
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- VMS diary booklet (Experimental)
  Interventions: Behavioral: VMS diary booklet
- Usual Care (e.g. Amsler grid monitoring) (Active Comparator)
  Interventions: Behavioral: Standard of Care

INTERVENTIONS:
Behavioral: VMS diary booklet
  Arms: VMS diary booklet
Behavioral: Standard of Care
  Arms: Usual Care (e.g. Amsler grid monitoring)

SUMMARY:
Exudative age-related macular degeneration ("wet" AMD) continues to be a leading cause of central vision loss in the US for those over fifty years of age, despite the availability of several effective interventions to contain damaging neovascularization (new, abnormal blood vessel growth). The effectiveness of treatments is challenged by patients' lack of ability to recognize the need for urgent care between regular office visits. The Amsler and Yanuzzi tests, the only widely used self-tests for AMD, have proven largely ineffective at enabling patients to recognize the signs that they should consult their retina specialist for treatment.

For optimal benefit, patients should be able to self-monitor their vision over time and detect changes that may be indicative of an exudative event. To facilitate compliance these observations should be part of a larger and more engaging program of AMD awareness and self-monitoring. Among the principal shortcomings of the current "gold-standard" Amsler grid are periodicity of the test pattern and lack of individual adjustment, and therefore the reliability and accuracy of this test are less than optimal for the detection of exudative retinal changes in AMD patients. In phase I of the current study, the investigatorsW developed and evaluated several versions of improved grids, both on paper and on the Internet. These patent-pending Visual and Memory Stimulating (VMS) grids proved at least equivalent to the Amsler grid in facilitating a substantial degree of recall of prior measurements, necessary for monitoring vision over time. Adjustment features were incorporated in the on-line version to allow patients to customize their grid to their particular visual field. In the phase II study the use of VMS grids will be supplemented by a test booklet that contains educational materials and diary based survey questions in addition to the printed VMS grids; the effectiveness of this booklet for self-monitoring will be compared the standard of care (Amsler grid).

Goal of the study is to demonstrate that use of the test booklet leads to more rapid identification of newly developing vision problems, earlier diagnosis and treatment of incipient wet AMD that should result in fewer people losing their vision and less severe losses of vision.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with a confirmed diagnosis of AREDS grade 3 or 4 AMD in at least one eye will be recruited for components 1 and 2 of the study. The participants will include healthy adults who are willing and able to complete the study tests. We will recruit AMD patients across a wide range of races and ages, but due to the prevalence of AMD, most of the patients will be Caucasian and over age 55. We will verify ocular diagnosis and visual function status of all subjects through records and communication provided by their retinal specialist.

Exclusion Criteria:

* Subjects with vision loss due to ocular pathology other than AMD or cataracts will be excluded.
* Subjects with cataract extraction in the last 3 months or capsulotomy in the last 24 hours in either eye will also be excluded, as well as those who are unable to give informed consent, non-English speaking or unable complete any other required study procedure.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 324 (Actual)
Dates: Start 2010-05-01 (Actual); Primary Completion 2015-03-26 (Actual); Study Completion 2015-03-26 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Johns Hopkins University Wilmer Eye Institute, Baltimore, Maryland, United States